CLINICAL TRIAL: NCT07002476
Title: A Prospective, Multicenter, Open-Label, Randomized Controlled Study of Early Intensive Lipid-Lowering in Endovascular Treatment for Acute Ischemic Stroke
Brief Title: Early Aggressive Strategy for Treatment of Lipid-Lowering in Acute Ischemic Stroke Delivered With Endovascular Therapy for Large Artery Occlusion
Acronym: EAST-LDL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-CVD-II-001
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: acute ischemic stroke; LDL-Cholersterol lowering; Endovascular Therapy; PCSK9; clinical trials
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Guideline-recommended standard of care
  Interventions: Drug: guideline-recommended SoC
- Investigational Group (Experimental): Guideline-recommended standard of care+intensive lipid-lowering therapy
  Interventions: Drug: Recaticimab (intensive)

INTERVENTIONS:
Drug: guideline-recommended SoC — Guideline-recommended SoC, including but not limited to oral lipid-lowering drugs, antiplatelet aggregation drugs, anticoagulant drugs, antihypertensive drugs, etc. It is to be determined by the investigator based on the subject's treatment needs.
  Arms: Control Group
Drug: Recaticimab (intensive) — Recaticimab is added to the guideline-recommended SoC. After randomization and before endovascular interventional treatment, patients will receive a subcutaneous injection of Recaticimab. The specific method is: Recaticimab 450 mg (3 vials) as a single subcutaneous injection, until the end of the follow-up for this study.
  Arms: Investigational Group

SUMMARY:
A prospective, multicenter, open-label, randomized controlled study to assess the effects of early intensive lipid-lowering initiated before endovascular treatment setting on (i) functional outcome in patients with acute ischemic stroke between preoperative intensive lipid-lowering therapy with PCSK9 inhibitor (PCSK9i) and guideline-recommended standard of care (SoC)(ii) safety in these patients.

DETAILED DESCRIPTION:
As a prospective, multicenter, open-label, randomized controlled clinical study, EAST-LDL will enroll 652 patients with acute ischemic stroke with anterior circulation large vessel occlusion undergoing endovascular treatment from approximately 10 clinical sites in China. This study aims to evaluate the effects of functional outcome according to an ordinal analysis of the full range of scores on the mRS, safety of lipid-lowering therapy, LDL-C goal attainment rate, change in inflammatory markers, incidence of recurrent ischemic stroke events , incidence of symptomatic intracranial hemorrhage transformation within 48 hours, incidence of new-onset hemorrhagic stroke, and incidence of MACEs in patients between early intensive lipid-lowering therapy with PCSK9 inhibitor and guideline-recommended standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older);
* Imaging diagnosis of acute ischemic stroke with anterior circulation large vessel occlusion (including: internal carotid artery, middle cerebral artery M1 and M2, anterior cerebral artery A1 and A2);
* Planned to undergo endovascular intervention within 24 hours of symptom onset (or last known well time) according to local guidelines;
* Provision of informed consent by the patient or his/her legally authorized representative (or by an appropriate agent according to local requirements).

Exclusion Criteria:

* ASPECTS score ≤5 on cranial CT imaging;
* Pre-existing functional impairment, with mRS score >2;
* Patients who are allergic to PCSK9 inhibitors;
* Patients who have received PCSK9 monoclonal antibody within 1 month prior to enrollment or PCSK9 siRNA therapy within 6 months prior to enrollment;
* Severe renal insufficiency, defined as estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73m2 at final screening;
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal;
* Severe, concomitant non-cardiovascular disease expected to reduce life expectancy to less than 3 months;
* Pregnant or lactating women;
* Patients who are participating in other clinical trials;
* Other conditions deemed unsuitable for inclusion in the clinical study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
favorable functional outcome (defined as an mRS score of 0-2) | Day 90
  the rate (%) of good functional outcome at 90 days (modified Rankin Scale [mRS] score 0-2). Modified Rankin Scale scores of 0 or 1 indicate good function without or with symptoms but not disability, score of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.

SECONDARY OUTCOMES:
mRS ordinal score | Day 90
  Modified Rankin Scale scores of 0 or 1 indicate good function without or with symptoms but not disability, score of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Change from baseline in NIHSS score | Day 14±3 days or before discharge
  0-42, higher scores indicates worse severity
Change from baseline in LDL-C | Day 14±3 days or before discharge
  Change from baseline in LDL-C at 14±3 days or before discharge
Change in inflammatory markers | Day 0, Day 14±3 days or before discharge
  Change from baseline in inflammatory markers at 14±3 days or before discharge;
Rate of severe disability(defined as mRS score of 3-5) | Day 90
  Modified Rankin Scale scores of 0 or 1 indicate good function without or with symptoms but not disability, score of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Incidence of recurrent ischemic stroke events | From enrollment to the end of treatment at 90 days
  Incidence of recurrent ischemic stroke events
Incidence of symptomatic intracranial hemorrhage transformation | Within 24-48 hours
  Incidence of symptomatic intracranial hemorrhage transformation within 24-48h;
Incidence of patients with new hemorrhagic stroke | From enrollment to 90 days
  Incidence of patients with new hemorrhagic stroke
Incidence of patients with major adverse cardiovascular events | From enrollment to 90 days
  Incidence of major adverse cardiovascular events (MACEs) within 90 days
Number of patients with serious adverse events | From enrollment to 90 days
  total number of serious adverse events reported during follow-up, according to standard definitions
Health related quality of life | Day 90
  according to the EQ-5D
NIHSS score | at 14±3 days or before discharge
  0-42, higher scores indicates worse severity
LDL-C goal attainment rate | at 14±3 days or before discharge
  LDL-C attained equal or lower than 1.8mmol/L or decrease by equal or more than 50%
Mortality rate | Day 90
  Death within 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai East Hospital, Study Chair — Tongji University
Locations (1):
- Shanghai East Hospital, Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT07002476/Prot_SAP_000.pdf